CLINICAL TRIAL: NCT03356613
Title: GenI: a Tool to Generate Paramedical Research Ideas
Acronym: GenI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: APPARA2016/GENI-KLEIN/ER
Record Dates: First submitted 2017-11-16; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Paramedical Staff Views of Research
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- focus group of paramedical staff from Nancy: During the focus group, the psychologist researcher asks the group a series of question about their views and opinions on research and how to make it.
  Interventions: Other: Focus group
- focus group of paramedical staff from Metz: During the focus group, the psychologist researcher asks the group a series of question about their views and opinions on research and how to make it.
  Interventions: Other: Focus group
- focus group of paramedical staff from Dijon: During the focus group, the psychologist researcher asks the group a series of question about their views and opinions on research and how to make it.
  Interventions: Other: Focus group
- focus group of paramedical staff from Bar-le-Duc: During the focus group, the psychologist researcher asks the group a series of question about their views and opinions on research and how to make it.
  Interventions: Other: Focus group
- Test of the tool by paramedical staff center 1: Paramedical staff who didn't participate to the focus group, will test the GenI tool to generate research ideas.
  Interventions: Other: test of the Geni tool
- Test of the tool by paramedical staff center 2: Paramedical staff who didn't participate to the focus group, will test the GenI tool to generate research ideas.
  Interventions: Other: test of the Geni tool

INTERVENTIONS:
Other: Focus group — An researcher in psychology will lead focus group on research views for paramedical staff
  Groups: focus group of paramedical staff from Bar-le-Duc; focus group of paramedical staff from Dijon; focus group of paramedical staff from Metz; focus group of paramedical staff from Nancy
Other: test of the Geni tool — The GenI tool built on paramedic's view will be tested.
  Groups: Test of the tool by paramedical staff center 1; Test of the tool by paramedical staff center 2

SUMMARY:
In order to develop paramedical research culture, the paramedical staff need adapted tools and methods. The GenI project (Research ideas generation) has for main objective the design and validation of a tool that will allow the identification of paramedical research ideas. This tool will be built based on paramedical staff views. Our hypothesis is that the use of the GenI tool will help to detect research ideas in paramedical health care that could lead to research projects.

ELIGIBILITY:
Inclusion Criteria:

* paramedical staff working in one of the 4 hospitals involved in the study

Exclusion Criteria:

* paramedical staff with a research degree
* paramedical staff that are paramedical coordinator in the hospital

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: paramedical staff
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the number of research ideas generated by a group of experts and by a group of paramedical staff | in 1 year
  At the end of each focus group, the group of paramedical staff and the group of experts will provide the list of ideas generated with or without the use of the tool. The number of ideas will be counted
Comparison of the pertinence of research ideas generated by a group of experts and by a group of paramedical staff | in 1 year
  Each research idea will be evaluated by an independent expert group on the "utility, innovation and feasibility" aspects (likert in 4 points) in order to compare the research ideas generated by paramedical groups (with the support of the GENI tool) and the research ideas generated by research experts groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Klein, Principal Investigator — CHRU Nancy Brabois
Locations (1):
- CIC 1433 Epidémiologie clinique, Vandœuvre-lès-Nancy, France